CLINICAL TRIAL: NCT02976181
Title: Registry to Improve the Adoption of Consensus Treatment Guideline (Brady MX)
Brief Title: Brady MX a Quality Improvement Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Brady MX
Record Dates: First submitted 2016-07-18; First posted 2016-11-29 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Sinus Node Disfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: IPG — Patient might require IPG device to be implanted under standard of care

SUMMARY:
Medtronic is sponsoring a quality improvement study called Brady MX. It is hypothesized that lack of awareness of treatment and diagnostics pathways result in lower number of referrals to implanters of IPG.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age
* Patient´s heart rate meets at least one of the following:

Patient has a sinus rate ≤ 50 OR a junctional escape rhythm no faster than 50 Patient has a history of exercise intolerance

* Patient complains of general fatigue, shortness of breath, shortness of breath with exertion, syncope, light headed dizziness, palpitations, lethargy, dyspnea OR malaise within the last 30 days that are not related to other discovered causes (such as untreated hypothyroidism or anemia)
* Patient (or patient´s legally authorized representative) is willing and able to sign and date written Patient Consent Form/Data Release Form

Exclusion Criteria:

* Patient has recent history of blood loss
* Patient has a medical history leading to suspicion of neurological disorder
* Patient has a history of Chronic Atrial Fibrilation
* Patient is enrolled or planing to participate in a concurrent drug and/or device study at any time during the course of this clinical study without documented pre-approval from Medtronic study manager
* Patient is not expected to survive 12 months
* Patient is anticipated to be unwilling or unable to comply with the clinical investigation plan

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bradycardia symptomatic patients
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Mexico (5):
  - Hospital General de Tijuana, Tijuana, Estado de Baja California
  - Hospital General de Cancun, Cancún, Quintana Roo
  - Hospital General del Estado de Sonora, Hermosillo, Sonora
  - Hospital Regional Universitario de Colima, Colima
  - Hospital General de Queretaro, Querétaro

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm/Group Observational Registry: Bradycardia patients with both signs and symptoms of bradycardia, prior to diagnosis of SND and IPG therapy
Period: Overall Study
Arm/Group | Single Arm/Group Observational Registry
Started | 113
Completed | 112
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm/Group Observational Registry
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean St. Dev. | 63.6 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 112
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 112
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.6 (4.9)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic Blood Pressure | 125.8 (20.7)
  Diastolic Blood Pressure | 74.9 (10.5)
Height [Mean (Standard Deviation); unit: cm] | 161.6 (9.1)
Weight [Mean (Standard Deviation); unit: kg] | 72.0 (13.8)
Symptoms [Count of Participants; unit: Participants]
  None | 6
  Chest pain | 17
  Dizziness / lightheadedness / presyncope | 63
  Dyspnea / shortness of breath | 30
  Edema | 4
  Exercise intolerance | 30
  Fatigue / weakness / lethargy | 35
  Malaise | 11
  Palpitations | 24
  Syncope | 25
Cardiac and Vascular History [Count of Participants; unit: Participants] — NYHA Classification: Stages of Heart Failure:
  Class I: No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    None | 40
    Brugada syndrome | 0
    Cardiac arrest | 0
    Cardiomyopathy | 1
    Congenital heart disease | 0
    Congestive heart failure | 2
    Coronary artery disease | 8
    Familial or inherited conditions with high risk fo | 0
    Hypertension | 55
    Hypotension | 1
    Left ventricular hypertrophy | 0
    Long Q/T Syndrome | 0
    Myocardial infarction | 6
    Primary / idiopathic electrical disease | 1
    Pulmonary hypertension (PH) | 0
    Valve dysfunction | 1
    Other cardiovascular history | 1
    Subject does not have heart failure | 29
    NYHA Class I | 53
    NYHA Class II | 12
    NYHA Class III | 1
    NYHA Class IV | 0
    No Cardiovascular Surgical History | 109
    Ablation | 0
    Carotid endarterectomy | 0
    Carotid stent | 0
    Coronary artery bypass graft (CABG) | 2
    Coronary artery intervention | 1
    Renal stent | 0
    Surgical MAZE | 0
    Valve repair | 0
    Valve replacement | 0
    No Atrial Arrythmias | 88
    Atrial asystole | 0
    AV nodal re-entrant tachycardia | 0
    Premature atrial complexes | 2
    Premature atrial complexes, non-conducted | 0
    SA nodal re-entry | 0
    Sinus node dysfunction | 20
    Atrial fibrillation, paroxysmal | 5
    Atrial fibrillation, persistant | 0
    Atrial fibrillation, permanent | 0
    Atrial flutter | 0
    Atrial tachycardia | 0
    Wandering atrial pacemaker | 0
    No Ventricular Arrhythmias | 107
    Idioventricular (ventricular escape) | 0
    Premature ventricular complexes (extrasystole) | 4
    Torsades de pointes | 0
    Ventricular asystole | 0
    Ventricular fibrillation | 0
    Ventricular flutter | 0
    Ventricular tachycardia | 1
    No AV Junctional Arrhythmias and Blocks | 104
    1st degree AV block | 3
    2nd degree AV block, type 1 (Wenckebach) | 0
    Other AV junctional arrhythmias and blocks | 4
    No Vascular History | 104
    Carotid artery disease | 0
    Cerebrovascular accident (stroke) | 3
    Deep vein thrombosis | 0
    Transient ischemic attack | 0
    Peripheral edema | 1
    Peripheral vascular disease | 1
    Poor peripheral perfusion | 0
    Pulmonary edema | 1
    Pulmonary embolism | 0
    Raynaud's phenomenon | 0
    Vascular aneurysm | 1
Endocrine History [Count of Participants; unit: Participants]
  None | 84
  Diabetes mellitus | 15
  Hormone replacement therapy | 0
  Hyperlipidemia | 4
  Hyperthyroidism | 2
  Hypothyroidism | 6
  Renal dysfunction, requiring dialysis | 1
  Renal dysfunction, not requiring dialysis | 6
  Renal dysfunction, unknown dialysis | 0
Respiratory / Pulmonary History [Count of Participants; unit: Participants]
  None | 105
  Asthma | 1
  Chronic obstructive pulmonary disease (COPD) | 3
  Emphysema | 0
  Hemoptysis | 0
  Lung cancer | 0
  Persistent cough | 1
  Pleural effusion | 0
  Pneumonia | 1
  Pulmonary fibrosis | 0
  Respiratory failure | 0
  Sleep apnea | 1
  Tuberculosis | 0
Smoking Status [Count of Participants; unit: Participants]
  Subject never smoked (habitually) | 60
  Subject currently smokes (habitually) | 13
  Subject has previously smoked (habitually) but doe | 38
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in the Proportion of Subjects Diagnosed With SND at Pre Specific Time.
Description: Because the study intervention was not conducted, it is not possible to compare the proportion of subjects with an SND diagnosis pre-intervention (Phase I) to the proportion post-intervention (Phase II). Instead, the proportion of subjects with an SND diagnosis in Phase I are reported
Time Frame: 6 and 12 months
Population: Number of SND Diagnoses by Time to Diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm/Group Observational Registry
Number analyzed (Participants) | 111
Participants
  6 Months | 69
  12 Months | 70

2. Secondary Outcome: Number of SND Subjects Receiving a Referral for an Indicated IPG Device After the Intervention
Description: The change between subjects referred to an indicated IPG will be measured after the intervention in total number of patients that are referred correctly.
  Because the study intervention was not conducted, it is not possible to compare the proportion of subjects receiving therapy referral for an indicated IPG pre-intervention (Phase I) to the proportion post-intervention (Phase II). Instead, the proportion of SND subjects receiving a referral for an indicated IPG device in Phase I are reported.
Time Frame: 3, 6, and 15 months
Population: Because the study intervention was not conducted, it is not possible to compare the proportion of subjects receiving indicated therapy pre-intervention (Phase I) to the proportion post-intervention (Phase II). Instead, the proportion of SND subjects receiving indicated IPG therapy in Phase I are reported
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm/Group Observational Registry: Bradycardia patients with both signs and symptoms of bradycardia, prior to diagnosis of SND and IPG therapy.
  Because the study intervention was not conducted, it is not possible to compare the proportion of subjects receiving indicated therapy pre-intervention (Phase I) to the proportion post-intervention (Phase II). Instead, the proportion of SND subjects receiving indicated therapy in Phase I are reported
Arm/Group | Single Arm/Group Observational Registry
Number analyzed (Participants) | 70
Participants
  3 Months | 17
  6 Months | 18
  15 Months | 19
  Not implanted | 51

ADVERSE EVENTS:
Time Frame: Adverse events were not collected in this study.
Description: Adverse events were not collected in this study.
Groups:
- Single Arm/Group Observational Registry: Bradycardia patients with both signs and symptoms of bradycardia, prior to diagnosis of SND and IPG therapy Adverse events were not collected in this study. There were no deaths reported in the study.
Arm/Group | Single Arm/Group Observational Registry
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No conclusions can be drawn from the amended analysis about whether educational interventions are able impact the clinical care pathway for bradycardia patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT02976181/Prot_SAP_000.pdf